CLINICAL TRIAL: NCT04398732
Title: Efficacy of Etanercept in Iraqi Patients With Moderate to Severe Psoriasis: 5 Years Data From Local Registry.
Brief Title: Study to Evaluate the Efficacy of Enbrel as a Biological Treatment in Moderate to Severe Plaque Psoriasis Patients
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801412
Record Dates: First submitted 2020-05-20; First posted 2020-05-21 (Actual); Results first posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-09

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients with moderate to severe plaque psoriasis: Iraqi patients diagnosed with moderate to severe plaque psoriasis that received Enbrel as treatment for disease.
  Interventions: Drug: Enbrel

INTERVENTIONS:
Drug: Enbrel — As provided in real world practice

SUMMARY:
This study is to evaluate available local data in Iraqi patients with moderate to severe psoriasis on Enbrel treatment with regards to efficacy, treatment regimen adherence and patient characterization (i.e. age, gender, smoking status) using data from the Dermatologists in Baghdad Teaching Hospital registry

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of moderate to severe plaque psoriasis receiving etanercept treatment for a minimum duration of 1 year.
* Age ≥18 years old.
* No history of using a biological treatment, other than etanercept, for treatment of moderate to severe plaque psoriasis or any other reason.

Exclusion Criteria:

* Etanercept use for treatment moderate to severe plaque psoriasis less than 1 year duration.
* Previous use of other biological treatments for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients data from the local registry at the Dermatology Center of Baghdad Teaching Hospital registry.
Sampling Method: Non-Probability Sample
Enrollment: 486 (Actual)
Dates: Start 2020-07-05 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1801412

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of Iraq's participants aged greater than or equal to (>=) 18 years, who received etanercept for at least 1 year for treatment of moderate to severe plaque psoriasis at dermatology center in the Baghdad teaching hospital were included in the study. Available data of maximum 5 years were evaluated in approximately 2.8 months of this retrospective, observational study.
Groups:
- Etanercept: Participants received etanercept to treat moderate-to-severe plaque psoriasis for at least 1 year under standard real world clinical practice. (In Iraq, the recommended dose of etanercept [Enbrel] is 25 milligrams [mg] administered twice weekly or 50 mg administered once weekly. Alternatively, 50 mg given twice weekly might be used for up to 12 weeks followed, if necessary, by a dose of 25 mg twice weekly or 50 mg once weekly). Data of these participants were studied for approximately 2.8 months in this study.
Period: Overall Study
Arm/Group | Etanercept
Started | 486
Completed | 436
Not Completed | 50
Not completed — Participants Who Did Not Meet Entrance Criteria | 50

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all participants whose data were included in this study for retrospective observation.
Groups:
- Etanercept: Participants received etanercept to treat moderate-to-severe plaque psoriasis for at least 1 year under standard real world clinical practice. (In Iraq, the recommended dose of etanercept [Enbrel] is 25 mg administered twice weekly or 50 mg administered once weekly. Alternatively, 50 mg given twice weekly might be used for up to 12 weeks followed, if necessary, by a dose of 25 mg twice weekly or 50 mg once weekly). Data of these participants were studied for approximately 2.8 months in this study.
Arm/Group | Etanercept
Number analyzed (Participants) | 486
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 240
  Male | 246
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Percent Body Surface Area (BSA) at Month 12
Description: Four body regions were evaluated: head and neck, upper limbs, trunk (including axillae and groin) and lower limbs (including buttocks). Scalp, palms and soles were excluded. BSA was calculated using handprint method. Number of handprints (size of participant's full palmer hand) fitting in affected area of a body region was counted. Maximum number of handprints were 10 for head and neck, 20 for upper limbs, 30 for trunk and 40 for lower limbs. Surface area of body region equivalent to 1 handprint: 1 handprint equal to (=) 10 percent (%) for head and neck, 5% for upper limbs, 3.33% for trunk and 2.5% for lower limbs. Percent BSA for a body region = total number of handprints in a body region * % surface area equivalent to 1 handprint. Overall % BSA for an individual: arithmetic mean of % BSA of all 4 body regions, ranged from 0 to 100%. Higher % BSA = greater severity of psoriasis.
Time Frame: Baseline, Month 12 (from the data retrieved and observed in approximately 2.8 months of this study)
Population: Analysis was performed on all participants whose data were included in this study for retrospective observation. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent BSA
Arm/Group | Etanercept
Number analyzed (Participants) | 422
Percent BSA | -21 (17.12191578)
Statistical Analysis 1: Comparison: Etanercept; Statistical analysis was performed on change from Baseline in percent BSA at Month 12; Test type: Other; p = 0.0001, Student's t-test

2. Primary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Month 12
Description: DLQI is a 10-item questionnaire that measures the impact of skin disease on participant's quality of life over the last week. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicated more impact on quality of life. Scores from all 10 questions added up to give DLQI total score range from 0 (not at all) to 30 (very much). Higher scores indicated more impact on quality of life of participants.
Time Frame: Baseline, Month 12 (from the data retrieved and observed in approximately 2.8 months of this study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 422
units on a scale | -17.2 (5.632051136)
Statistical Analysis 1: Comparison: Etanercept; Statistical analysis was performed on change from baseline in DLQI at Month 12; Test type: Other; p = 0.0001, Student's t-test

3. Primary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Score at Month 12
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and the "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 (no disease) to 72.0 (maximum disease), with higher scores representing greater severity of psoriasis.
Time Frame: Baseline, Month 12 (from the data retrieved and observed in approximately 2.8 months of this study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 422
units on a scale | -16.44 (9.062008607)
Statistical Analysis 1: Comparison: Etanercept; Statistical analysis was performed on change from baseline in PASI at Month 12; Test type: Other; p = 0.0001, Student's t-test

4. Secondary Outcome: Percent Body Surface Area (BSA) at Baseline, Month 4, and Month 12 in Participants Adherent and Not Adherent to Treatment
Description: Four body regions were evaluated: head and neck, upper limbs, trunk (including axillae and groin) and lower limbs (including buttocks). Scalp, palms and soles were excluded. BSA was calculated using handprint method. Number of handprints (size of participant's full palmer hand) fitting in affected area of body region was counted. Maximum number of handprints were 10 for head and neck,20 for upper limbs,30 for trunk and 40 for lower limbs. Surface area of body region equivalent to 1 handprint: 1 handprint = 10% for head and neck, 5% for upper limbs, 3.33% for trunk and 2.5% for lower limbs. % BSA for body region=total number of handprints in a body region * % surface area equivalent to 1 handprint. Overall % BSA for individual: arithmetic mean of % BSA of all 4 body regions, ranged from 0 to 100%. Higher % BSA=greater severity of psoriasis. This outcome measure evaluated comparison in % BSA between participants adherent and not adherent to treatment at Baseline, Month 4 and 12.
Time Frame: Baseline, Month 4 and Month 12 (from the data retrieved and observed in approximately 2.8 months of this study)
Population: Analysis was performed on all participants whose data were included in this study for retrospective observation. Here, "Number Analyzed" signifies participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: Percent BSA
Groups:
- Etanercept: Participants Adherent to Treatment: Participants received etanercept to treat moderate-to-severe plaque psoriasis for at least 1 year under standard real world clinical practice and were adherent to treatment. (In Iraq, the recommended dose of etanercept [Enbrel] is 25 mg administered twice weekly or 50 mg administered once weekly. Alternatively, 50 mg given twice weekly might be used for up to 12 weeks followed, if necessary, by a dose of 25 mg twice weekly or 50 mg once weekly). Data of these participants were studied for approximately 2.8 months in this study.
- Etanercept: Participants Not Adherent to Treatment: Participants received etanercept to treat moderate-to-severe plaque psoriasis for at least 1 year under standard real clinical practice and were not adherent to treatment. (In Iraq, the recommended dose of etanercept [Enbrel] is 25 mg administered twice weekly or 50 mg administered once weekly. Alternatively, 50 mg given twice weekly might be used for up to 12 weeks followed, if necessary, by a dose of 25 mg twice weekly or 50 mg once weekly). Data of these participants were studied for approximately 2.8 months in this study.
Arm/Group | Etanercept: Participants Adherent to Treatment | Etanercept: Participants Not Adherent to Treatment
Number analyzed (Participants) | 417 | 69
Percent BSA
  Baseline | 27.56 (19.030) | 32.84 (21.324)
  Month 4: number analyzed (Participants) | 413 | 69
  Month 4 | 20.1 (11.7) | 31.7 (21.8)
  Month 12: number analyzed (Participants) | 353 | 69
  Month 12 | 8.7 (6.8) | 11.1 (8.9)
Statistical Analysis 1: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Baseline; Test type: Other; p = 0.036, Student's t-test
Statistical Analysis 2: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Month 4; Test type: Other; p = 0.0001, Student's t-test
Statistical Analysis 3: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Month 12; Test type: Other; p = 0.0001, Student's t-test

5. Secondary Outcome: Dermatology Life Quality Index (DLQI) Score at Baseline, Month 4 and Month 12 in Participants Adherent and Not Adherent to Treatment
Description: DLQI is a 10-item questionnaire that measures the impact of skin disease on participant's quality of life over the last week. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicated more impact on quality of life. Scores from all 10 questions added up to give DLQI total score range from 0 (not at all) to 30 (very much). Higher scores indicated more impact on quality of life of participants. This outcome measure evaluated comparison in DLQI score between participants adherent and not adherent to treatment at Baseline, Month 4 and 12.
Time Frame: Baseline, Month 4 and Month 12 (from the data retrieved and observed in approximately 2.8 months of this study)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept: Participants Adherent to Treatment | Etanercept: Participants Not Adherent to Treatment
Number analyzed (Participants) | 417 | 69
units on a scale
  Baseline | 24.50 (4.438) | 24.94 (2.838)
  Month 4: number analyzed (Participants) | 413 | 69
  Month 4 | 16.6 (6.3) | 21.1 (6.8)
  Month 12: number analyzed (Participants) | 353 | 69
  Month 12 | 6.6 (4.5) | 11.3 (7.2)
Statistical Analysis 1: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Baseline; Test type: Other; p = 0.42, Student's t-test
Statistical Analysis 2: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Month 4; Test type: Other; p = 0.0001, Student's t-test
Statistical Analysis 3: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Month 12; Test type: Other; p = 0.0001, Student's t-test

6. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Score at Baseline, Month 4 and Month 12 in Participants Adherent and Not Adherent to Treatment
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and the "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 (no disease) to 72.0 (maximum disease), with higher scores representing greater severity of psoriasis. This outcome measure evaluated comparison in PASI score between participants adherent and not adherent to treatment at Baseline, Month 4 and 12.
Time Frame: Baseline, Month 4 and Month 12 (from the data retrieved and observed in approximately 2.8 months of this study)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept: Participants Adherent to Treatment | Etanercept: Participants Not Adherent to Treatment
Number analyzed (Participants) | 417 | 69
units on a scale
  Baseline | 21.980 (10.0055) | 22.458 (12.6765)
  Month 4: number analyzed (Participants) | 413 | 69
  Month 4 | 14.5 (8.8) | 21.7 (15.8)
  Month 12: number analyzed (Participants) | 353 | 69
  Month 12 | 4.8 (3.9) | 9.7 (6.4)
Statistical Analysis 1: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Baseline; Test type: Other; p = 0.72, Student's t-test
Statistical Analysis 2: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Month 4; Test type: Other; p = 0.0001, Student's t-test
Statistical Analysis 3: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Month 12; Test type: Other; p = 0.0001, Student's t-test

7. Other Pre Specified Outcome: Change From Baseline in Percent Body Surface Area (BSA) at Month 4
Description: Four body regions were evaluated: head and neck, upper limbs, trunk (including axillae and groin) and lower limbs (including buttocks). Scalp, palms and soles were excluded. BSA was calculated using handprint method. Number of handprints (size of participant's full palmer hand) fitting in affected area of a body region was counted. Maximum number of handprints were 10 for head and neck, 20 for upper limbs, 30 for trunk and 40 for lower limbs. Surface area of body region equivalent to 1 handprint: 1 handprint = 10 % for head and neck, 5% for upper limbs, 3.33% for trunk and 2.5% for lower limbs. Percent BSA for a body region = total number of handprints in a body region * % surface area equivalent to 1 handprint. Overall % BSA for an individual: arithmetic mean of % BSA of all 4 body regions, ranged from 0 to 100%. Higher % BSA = greater severity of psoriasis.
Time Frame: Baseline, Month 4 (from the data retrieved and observed in approximately 2.8 months of this study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent BSA
Arm/Group | Etanercept
Number analyzed (Participants) | 482
Percent BSA | -6.8 (17.39310208)
Statistical Analysis 1: Comparison: Etanercept; Statistical analysis was performed on change from Baseline in percent BSA at Month 4; Test type: Other; p = 0.0001, Student's t-test

8. Other Pre Specified Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Month 4
Description: as for outcome 2
Time Frame: Baseline, Month 4 (from the data retrieved and observed in approximately 2.8 months of this study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 482
units on a scale | -7.3 (5.70876519)
Statistical Analysis 1: Comparison: Etanercept; Statistical analysis was performed on change from baseline in DLQI at Month 4; Test type: Other; p = 0.0001, Student's t-test

9. Other Pre Specified Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Score at Month 4
Description: as for outcome 3
Time Frame: Baseline, Month 4 (from the data retrieved and observed in approximately 2.8 months of this study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept
Number analyzed (Participants) | 482
units on a scale | -6.64 (10.35036231)
Statistical Analysis 1: Comparison: Etanercept; Statistical analysis was performed on change from baseline in PASI at Month 4; Test type: Other; p = 0.0001, Student's t-test

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not collected for the study
Description: Due to non-interventional nature of study, the minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) could not meet, hence adverse events were not collected and reported.
Arm/Group | Etanercept
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT04398732/Prot_SAP_000.pdf